CLINICAL TRIAL: NCT05647993
Title: Comparing of Cefazolin Plus Azithromycin Versus Cefazolin Alone in Prevention of Febrile Morbidity After Emergency Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Comparing of Cefazolin Plus Azithromycin Versus Cefazolin in Prevention of Febrile Morbidity After Emergency Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 65094
Record Dates: First submitted 2022-11-04; First posted 2022-12-13 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-02

CONDITIONS: Febrile Morbidity After Emergency Cesarean Section
MeSH Terms: interventions — Azithromycin; Cefazolin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo) (Placebo Comparator): Patient will receive standard antimicrobial prophylaxis(cefazolin intravenously weight dependent) and placebo(0.9% NaCl 100 ml intravenously) before the incision
  Interventions: Drug: Cefazolin; Drug: Sodium Chloride 0.9% Intravenous Solution
- azithromycin (Experimental): Patient will receive standard antimicrobial prophylaxis(cefazolin intravenously weight dependent) and azithromycin 500 mg intravenously before the incision
  Interventions: Drug: Azithromycin Injection [Zithromax]; Drug: Cefazolin

INTERVENTIONS:
Drug: Azithromycin Injection [Zithromax] — Intervention group patient will receive standard antimicrobial prophylaxis(cefazolin intravenously weight dependent) and azithromycin 500 mg intravenously before the incision
  Other Names: azithromycin
  Arms: azithromycin
Drug: Cefazolin — All the participants will receive the cefazolin intravenously. The dosage of the cefazolin is depend on participant's weight. The participant with weight less than 80kg will receive cefazolin 1 gm and between 80-120kg will receive cefazolin 2 gm and for the participant with more than 120kg will receive cefazolin 3 gm before the incision.
  Other Names: azithromycin; placebo comparator
Drug: Sodium Chloride 0.9% Intravenous Solution — For the placebo group will receive the cefazolin intravenously and 0.9% NaCl 100ml before the incision
  Other Names: placebo comparator
  Arms: Control group (Placebo)

SUMMARY:
Cesarean section is the common surgery in world wide. But the complication like febrile morbidity such as surgical site infection, fever, urinary tract infection and endometritis can be occurred even giving the standard antibiotics. Therefore if wider bacterial spectrum coverage antibiotic like azithromycin is added to the standard antimicrobial prophylaxis(1st generation cephalosporin), the incidence of febrile morbidity could be reduced. We will compare the regimen of cefazolin plus azithromycin and standard regimen of cefazolin alone in prevention of febrile morbidity after emergency cesarean section.

DETAILED DESCRIPTION:
This study was designed to evaluate the effect of azithromycin on the incidence of febrile morbidity after the emergency cesarean section. The standard antimicrobial prophylaxis which is recommended by the ACOG is the 1st generation cephalosporin intravenously only but some of the bacteria that can cause the febrile morbidity after cesarean section wouldn't be killed by the 1st generation cephalosporin. The antibiotic that can cover them is macrolide group antibiotic such as azithromycin. Therefore this study will compare the regimen of standard antimicrobial prophylaxis and the regimen of standard antimicrobial prophylaxis with azithromycin intravenously in preventing the febrile morbidity after emergency cesarean section. Control group will receive the 1st generation cephalosporin intravenously and the intervention group will receive the 1st generation cephalosporin with azithromycin 500mg intravenously. Primary outcome is febrile morbidity which assessed at postoperative day 3. The definition of the febrile morbidity in this study is including surgical site infection, endometritis, urinary tract infection and fever alone. Secondary outcomes are febrile morbidity at postoperative day 7 and day30, neonatal outcome and adverse effect from azithromycin use.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy with a gestation of 24 weeks or more
2. Undergoing non-elective cesarean delivery during labor or rupture of membrane more than 4 hr
3. No allergy to macrolide such as azithromycin and clindamycin
4. Provide informed consent
5. Partner of participant allows the patient to participate the research

Exclusion Criteria:

1. Use of azithromycin within 7 days before enrollment
2. Chorioamnionitis or other infection requiring postpartum antibiotic therapy (except for antibiotics for group B streptococcus)
3. Liver disease (Cirrhosis or AST more than 3 times the upper normal limit)
4. Serum creatinine level of more than 2.0 mg/dL or need dialysis
5. Diarrhea at the time of enrollment
6. Maternal heart disease
7. Use of medication known to prolonged the QT interval

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — for singleton pregnant
Enrollment: 172 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of febrile morbidity at postoperative day 3 | postoperative day 3
  Patient will be assessed at postoperative day 3. Febrile morbidity is including surgical site infection, endometritis, urinary tract infection and fever. There is the questionnaire for the assessor to check if there is the febrile morbidity or not. (There are criteria diagnosis of febrile morbidity from the CDC in the questionnaire)

SECONDARY OUTCOMES:
adverse drug effect | baseline and postoperative day 3, 7 and 30
  Any adverse drug effect of azithromycin such as diarrhea, urticaria, and anaphylactic shock
Incidence of adverse Neonatal outcome | baseline and postoperative day 3, 7 and 30
  any adverse neonatal outcome such as NICU admission, neonatal sepsis, need phototherapy, respiratory distress, Apgar score, neonatal death and neonatal enterocolitis (Assessed and diagnosis by pediatric doctor)
Incidence of febrile morbidity at postoperative day 7 and day 30 | postoperative day 7 and day 30
  Patient will be assessed at postoperative day 7 and day 30. Febrile morbidity is including surgical site infection, endometritis, urinary tract infection and fever. There is the questionnaire for the assessor to check if there is the febrile morbidity or not. (There are criteria diagnosis of febrile morbidity from the CDC in the questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No